CLINICAL TRIAL: NCT03686592
Title: Psychological Effect of the pancréatectomy: a Feeling of Strangeness
Acronym: REPPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REPPSE-IPC 2017-007
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Pancreatectomy
Keywords: Pancreatic cancer; body awareness; post-traumatic stress
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pancreatectomized patients (Experimental): Patients with pancreatic cancer who underwent a pancreatectomy at Institut Paoli Calmettes
  Interventions: Other: Measurement of body awareness
- Volunteers (Active Comparator)
  Interventions: Other: Measurement of body awareness

INTERVENTIONS:
Other: Measurement of body awareness — Questionnaires+ interviews

SUMMARY:
The cancer of the pancreas represents 1,8 % of cancers in France, with 9040 new cases in 2011 (France). This cancer is known to be of dark forecast. Indeed, of late clinical expression, is diagnosed most of the time at a late stage . For that reason, the cancer of the pancreas is considered as the one who presents the least good prognosis for survival. He affects more frequently the men than the women (rate of incidence of 7,7 against 4,7 cases for 100 000). Between 1980 and 2005, the incidence increased by 3,8 % at the women, by 2,0 % at the men (INCA Source, on 2012). The number of cases of cancer of the pancreas in the world is estimated at 278 684, with 266 669 deaths a year (Cancer Incidence and Mortality Worldwide - Globocan, on 2008).

In these cases of very grave cancers, the surgery represents the unique treatment to curative aim, although always not warning of a risk of relapse, and susceptible of entrainer to complications. Thus the pancréatectomy establishes a modality of specific treatment. Remaining the ultimate chance of cure, it is only rarely possible. Indeed, only 10 in 20 % of the cancers of the pancreas exocrines can be handled by surgery when the latter establish 95 % of the cases of pancreatic cancer.

To date, the psychosomatic approach goes away from the search for the causes to be interested more and more in the psychological consequences of the somatic disorders, what we wish to study in the present search.

Once the surgical indication was put, one of the key elements in the psychological plan is the uncertainty as for the outcome of the ablation, as well as the consequences psychopathologiques which ensue from it. The mutilation of an organ, whatever it is, can have an impact on the identity of the person constituting at the same time a physical and narcissistic wound, while having psychological effect at the sick person such as of the anxiety, a depression, or another a state of post-traumatic stress.

More exactly, a study was able to show a positive relation between cancer of the pancreas and depression in a retrospective study. A review of literature concerning the specific relations between depression and cancer of the pancreas was also realized. Besides, 50 % of the patients have a significant level of anxiety and 15 % of depression. A study was nevertheless able to bring to light that the depression does not affect the survival of the patient. Finally, a study was also able to find a decrease marked with the quality of life of the patients during the next first 6 months the operation.

Various studies so studied the quality of life of the patients reached of a cancer of the pancreas in particular in comment surgery. It is also advisable to specify that besides the depression and the quality of life, the strategies of adaptation of the patients having undergone a pancréatectomy were also the object of studies. However, none documented, to date, the specific psychological consequences described clinically by certain patients, in particular the feeling of confusion and strangeness felt, and it in association with the possible presence of a state of post-traumatic stress in several weeks of the operation.

DETAILED DESCRIPTION:
The objective of this exploratory research is to identify and to describe the psychological specificities of the pancréatectomy which can in particular include the feeling of strangeness and confusion at the sick person towards its own body.

It will also be a question of estimating the relations of this experience with a possible state of post-traumatic stress. Indeed, the announcement of the cancer as well as the surgery in itself are two elements which can be considered as traumatic.

For it a double methodology will be used, with a design cross-sectionnal: a quantitative shutter(sector) (auto-questionnaires) allowing to study aspects of the psychosocial functioning, and qualitative shutter with a semi-structured interview concerning the subjective experience of the participants. For the interpretation of the meditative data of the conversations, we shall use the phenomenological interpretative analysis ( IPA) which will allow us to investigate in a comprehensive way the subjective experience of the participants by studying the way the people give meaning to the fact that they live.

ELIGIBILITY:
Inclusion Criteria:

* Patient of at least 18 years, presenting a good understanding and a practice of the French language,
* Having undergone a pancreatectomy (pancreatic cancer),
* Signed Consent of participation,
* Affiliating to a national social security or beneficiary of such regimen

Exclusion Criteria:

* Other medical or psychiatric affection,
* Level of incompatible cognitive efficiency with the answer to auto-questionnaires,
* Patient in emergency situation, major person being the object of a legal protective measure (major under guardianship, guardianship or protection(saving) of justice), or outside state to express its consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Measurement of body awareness | 1 day
  body awareness will be measured thanks to a scale of Body Connection questionnaire

SECONDARY OUTCOMES:
Evaluation of post-traumatic stress | 1 day
  Post-traumatic stress will be evaluated thanks to a questionnaire+ an interview

CONTACTS AND LOCATIONS:
Locations (1):
- GENRE, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut Paoli-Calmettes — http://institutpaolicalmettes.fr